CLINICAL TRIAL: NCT03509584
Title: Phase I Multicenter Trial Combining Nivolumab, Alone or With Ipilimumab, Plus Hypo-fractionated Radiotherapy for Pretreated Advanced Stage Non-small Cell Lung Cancer Patients
Brief Title: Phase I Multicenter Trial Combining Nivolumab, Ipilimumab and Hypo-fractionated Radiotherapy for Pretreated Advanced Stage Non-small Cell Lung Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: SAFETY
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-21; 2017-001198-18 (EudraCT Number)
Record Dates: First submitted 2018-04-10; First posted 2018-04-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiation Dose Hypofractionation; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- part #1a (Experimental): non-small cell lung cancer (NSCLC) patients with bone metatase(s) eligible for localized hypo-fractionated radiotherapy
  Interventions: Radiation: hypofractionated radiotherapy; Drug: nivolumab
- part #1b (Experimental): non-small cell lung cancer (NSCLC) patients with bone metatase(s) eligible for localized hypo-fractionated radiotherapy
  Interventions: Radiation: hypofractionated radiotherapy; Drug: nivolumab; Drug: Ipilimumab
- part #2a (Experimental): NSCLC patients eligible for a localized radiotherapy of one target lesion (outside the brain)
  Interventions: Radiation: hypofractionated radiotherapy; Drug: nivolumab
- part #2b (Experimental): NSCLC patients eligible for a localized radiotherapy of one target lesion (outside the brain)
  Interventions: Radiation: hypofractionated radiotherapy; Drug: nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Radiation: hypofractionated radiotherapy — Stereotactic hypo-fractionated irradiation (3 x 8 Gys) radiotherapy fraction
Drug: nivolumab — administration of nivolumab
Drug: Ipilimumab — administration of ipilimumab
  Arms: part #1b; part #2b

SUMMARY:
Nivolumab is superior to docetaxel monotherapy as second line treatment in advanced stage non-small cell lung cancer (NSCLC) patients. However, the long term survival advantage seems to be limited to a 20% proportion of treated patients. To date, no definitive biomarker, including tumor cells or infiltrative cells PD-L1 expression, has been demonstrated to predict nivolumab (or other PD1 or PD-L1 inhibitors) efficacy. Ipilimumab has also suggested efficacy in the same patient population. Finally, the addition of ipilimumab to nivolumab has a suggested better efficacy over nivolumab alone in advanced stage NSCLC patients with an acceptable safety profile.

In parallel, hypo-fractionated radiotherapy alone has been suggested to elicit the immune system activity as demonstrated by the occurrence of an abscopal effect. Some case reports in melanoma but also lung cancer patients reinforced this hypothesis.

Furthermore, preclinical and clinical data suggest that radiation may have a synergistic effect with antibodies targeting the immune checkpoints (PD1, PD-L1, CTLA4) and improve antitumor efficacy. Moreover, it has been shown that fractionated radiotherapy delivered in combination with aPD-1 or aPD-L1 mAbs is able to generate efficacious CD8þ T-cell responses that will in turn improve local tumor control, long-term survival, and protection against tumor rechallenge.

Therefore, the combination of single fraction or hypo-fractionated radiotherapy with the anti PD1 nivolumab and/or the anti CTLA4 ipilimumab warrants further investigation. However, a large number of doses, sequences and schedules remain possible. In order to select the best combination, a mathematical modeling of immunotherapy in cancer and its synergy with radiotherapy has been set up. This work provides with mathematical formulas to link the drug serum concentrations of nivolumab and ipilimumab, and the dose of radiation therapy, to the immune response. In silico, the single and three fractions schedule have been found to have the same efficacy while activation of the immune response seems to be better using a hypo-fractionated (less than 6 fractions) radiotherapy in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC
* One site of measureable disease by RECIST 1.1
* Eligible for localized palliative radiotherapy of a bone lesion as per current national and international recommendations (part #1) or
* Ability to tolerate hypo-fractionated radiotherapy of a tumoral lesion chosen according to the lower risk of radiation adverse event (lymph node > subcutaneous > liver > bone > lung) (part #2)
* Received at least one prior line of therapy for incurable or metastatic NSCLC
* Disease progression at study entry

Exclusion Criteria:

* Received systemic anticancer therapy within the previous 21 days
* Human immunodeficiency virus (HIV), hepatitis B or C, or severe/uncontrolled infections or concurrent illness, unrelated to the tumor, requiring active therapy
* Any condition requiring concurrent systemic immunosuppressive therapy
* Known immunodeficiency disorders, either primary or acquired
* Bone lesion with indication of surgery (part #1) ; especially in case of spinal compression.
* Known leptomeningeal disease
* Active malignancies within 12 months with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* Prior treatment with immune checkpoints inhibitors
* Administration of a live, attenuated vaccine within 30 days prior to first dose of study drug
* Long-term use of systemic corticosteroids (unless to a dose of 20mg of methylprednisolone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Incidence of immune related adverse events | 48 weeks
  evaluate the safety of the combination of the radiotherapy plus nivolumab alone or in combination with ipilimumab, by physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France